CLINICAL TRIAL: NCT03718611
Title: A Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of Oral Administration of BR9001 Compared With BR900A in Healthy Subjects
Brief Title: To Evaluate the Pharmacokinetics and Safety of Oral Administration of BR9001 Compared With BR900A in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BR-TFD-CT-101
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Generic
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): BR900A - Wash out - BR9001
  Interventions: Drug: BR9001; Drug: BR900A
- Sequence 2 (Experimental): BR9001 - Wash out - BR900A
  Interventions: Drug: BR9001; Drug: BR900A

INTERVENTIONS:
Drug: BR9001 — BR9001 is a test drug as generic
Drug: BR900A — BR900A is a reference drug

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of oral administration of BR9001 compared with BR900A in healthy subjects

DETAILED DESCRIPTION:
This is an open-label, randomized, crossover study to evaluate the pharmacokinetics and safety. Within each period, randomized subjects will be take 2 dosing regimens that BR9001 or BR900A.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19-50 years of age
* Body mass index (BMI) ≥ 18.5 and ≤ 27.0 kg/m^2 at screening
* Medically healthy with no clinically significant medical history
* No clinically significant result with laboratory test including chemistry, serum, urine test within 3 weeks in prior to administration of investigational product
* Understands the study procedures in the Informed consent form (ICF), and be willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Creatinint clearance < 80 mL/min (using Cockcroft-Gault) at screening.
* Whole blood donation within a 2 months prior to the first dose of study drug.
* Participation in another clinical trial or bioequivalence study within 12 weeks prior to the first dose of study drug(s).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-24 hours after administration
  Maximum concentration of drug in plasma of BR9001 and BR900A
AUClast | 0-24 hours after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 to the last observed plasma concentration of BR9001 and BR900A

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D. PhD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No